CLINICAL TRIAL: NCT02022527
Title: Cost Effectiveness Analysis for Combination Of Aspirin And Warfarin Versus Warfarin Alone In Egyptian Patients With Heart Valve Prosthesis
Brief Title: Cost Effectiveness Analysis In Patients With Heart Valve Prosthesis
Acronym: HVP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmacoeconomic Unit, Egypt (Other Government)
Responsible Party: Principal Investigator, Gihan Hamdy Elsisi, Head of Pharmacoeconomic Unit, Pharmacoeconomic Unit, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEU2013
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Complications Due to Heart Valve Prosthesis
Keywords: Cost-Effectiveness,; Heart valve prosthesis; Warfarin,; Aspirin,; Egypt
MeSH Terms: interventions — Aspirin; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination (Experimental): Warfarin tablets adjusted according to international normalized ratio (INR) (2 for Aortic Valve Replacement & 2.5-3 for Mitral Valve Replacement, 2.5-3.5 for Double Valve Replacement) and oral 75 mg Acetyl Salicylic Acid tablets daily long life.
  Interventions: Drug: Acetyl Salicylic Acid; Drug: Warfarin
- Warfarin (Active Comparator): Warfarin tablets adjusted according to INR (2 for Aortic Valve Replacement & 2.5-3 for Mitral Valve Replacement, 2.5-3.5 for Double Valve Replacement) and placebo long life.
  Interventions: Drug: Warfarin; Drug: Placebo (for Aspirin)

INTERVENTIONS:
Drug: Acetyl Salicylic Acid
  Other Names: Aspirin
  Arms: Combination
Drug: Warfarin
  Other Names: Marevan
Drug: Placebo (for Aspirin) — Sugar pill manufactured to mimic 75 mg Aspirin
  Arms: Warfarin

SUMMARY:
The combined Antiplatelet and Anticoagulant treatment decreased thrombus formation and overall mortality. Also the initiation of an efficacious early anticoagulation protocol is important because of its potential impact on the rate of early thromboembolic complications after mechanical valve implantation. An important question that remains to be answered is whether the combination would be cost effective than Warfarin alone, with a reduction in major bleeding. In addition, the knowledge about its cost-effectiveness has not yet been established in Egypt. The aim of this trial based economic evaluation is to conduct a cost-effectiveness analysis for combination of low-dose Aspirin and Warfarin versus Warfarin alone in prosthetic valve patients from the medical provider perspective specially that a misconception is still existed between the physicians in Egypt that the cost of complications is not worthy so our main aim is to test the cost of complications.

DETAILED DESCRIPTION:
The measurements will be assessed:

A- Number of patients improved during follow up:

1. Demographic data
2. Diagnosis
3. Laboratory tests (CBC, Prothrombin Time, liver and renal function tests)
4. Echocardiography profile

B-Costs:

Direct medical costs will be assessed directly from hospital's records and tender lists.

ELIGIBILITY:
Inclusion Criteria:

Patients operated in Ain Shams University Hospitals for aortic and/ or mitral valve replacement.

Exclusion Criteria:

* Congenital blood disorders, Hemophilia.
* Advanced liver disease
* Advanced renal disease (dialysis patients)
* Aspirin sensitivity
* Autoimmune diseases
* Biological bioprosthesis valves
* Non-compliant & Drop out patient
* Pregnant women
* Caucasians.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Valve Thrombosis | one year

SECONDARY OUTCOMES:
Major Systemic Embolism, | one year
Non-fatal intracranial hemorrhage | one year
Major extra cranial hemorrhage, | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gihan H Elsisi, Msc, Principal Investigator — Pharmacoeconomic Unit; Manal H Elhamamsy, PhD, Study Chair — Faculty of pharmacy, Ain Shams University; Mohamed ME Mazar, PhD, Study Director — Central Administration for Pharmaceutical Affairs
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

REFERENCES:
- [Background] Mohamed H. Antithrombotic therapy in patients with prosthetic heart valves. Libyan J Med. 2009 Mar 1;4(1):54-6. doi: 10.4176/090115. PMID 21483507